CLINICAL TRIAL: NCT00048295
Title: ISIS 2302-CS21, Phase 3 Double-Masked, Placebo-Controlled Study of Alicaforsen (ISIS 2302), an Antisense Inhibitor of ICAM-1, for the Treatment of Patients With Active Crohn's Disease
Brief Title: Alicaforsen (ISIS 2302) in Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 2302-CS21
Record Dates: First submitted 2002-10-29; First posted 2002-10-30 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — alicaforsen

INTERVENTIONS:
Drug: Alicaforsen

SUMMARY:
ISIS 2302 is an antisense oligonucleotide drug that reduces the production of a specific protein called intercellular adhesion molecule (ICAM-1), a substance that plays a significant role in the increase of inflammation. People with Crohn's disease have been shown to over-produce ICAM-1 in their gut tissues. Alicaforsen works by blocking ICAM-1 messenger RNA, the "instruction" molecule that is required for the production of ICAM-1 protein. This trial will examine effects of alicaforsen delivered by 2-hour intravenous infusion over a four-week period, compared to a placebo. Patients may remain on stable background 5-ASA, antibiotic, or immunosuppressive drugs, and prednisone (or equivalent) at </= 30 mg per day.

ELIGIBILITY:
Inclusion Criteria

1. Age >/= 12 years
2. Weight >/= 36 kg
3. CDAI score of 220 - 400
4. Documentation of Crohn's disease activity by endoscopy, biopsy or imaging in the last 2 years
5. No TNF-α inhibitor treatment for three months prior to first study drug infusion

Exclusion Criteria

1. Known severe, fixed, symptomatic stenosis of the small or large intestine with significant dilation
2. Extensive external fistulization (> 3 external fistulae which are expressible with gentle compression); colostomy or ileostomy
3. Active infection, including infectious colitis, or infection with HIV, Hepatitis B or Hepatitis C
4. Malignancy within 3 years or poorly controlled medical illness
5. Requires intravenous heparin therapy or with a history of a bleeding problem

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (2):
  - Kortrijk
  - Roeselare
- Czechia (4):
  - Hradic Kralove 2
  - Olomouc
  - Prague
  - Ústí nad Orlicí
- Germany (2):
  - Minden
  - Münster
- Torino, Italy
- Poland (4):
  - Krakow
  - Szczecin
  - Warsaw
  - Wroclaw
- Spain (2):
  - Barcelona
  - Valencia

REFERENCES:
- See also: Type "ISIS 2302" in search box — http://www.centerwatch.com
- See also: Type "ISIS 2302" in search box, then click on "Crohn's Disease Alicaforsen Investigation" — http://www.acurian.com